CLINICAL TRIAL: NCT00922766
Title: Effectiveness And Safety Of Dalteparin In Patients With Acute Coronary Syndromes Without ST Elevations In Clinical Practice
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6301088
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Results first posted 2011-11-11 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Acute Coronary Syndrome
Keywords: dalteparin non-ST segment elevated acute coronary syndromes
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Dalteparin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1.0
  Interventions: Drug: Dalteparin

INTERVENTIONS:
Drug: Dalteparin — Patients prescribed dalteparin for non-ST segment elevated acute coronary syndromes in nursing home patients who will be treated conservatively (without corornary intervention [PCI] or coronary artery bypass graft [CABG] within 48 hours).

SUMMARY:
To collect data on safety and effectiveness of dalteparin in the management of non-ST segment elevated acute coronary syndromes in nursing home patients who will be treated conservatively (without percutaneous corornary intervention [PCI] or coronary artery bypass graft [CABG] within 48 hours).

DETAILED DESCRIPTION:
t

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of 18 years or more presenting with chest pain will be potentially eligible for inclusion in the study if they satisfy the criteria for unstable coronary artery disease per the investigator's routine practice and have received at least one injection of Fragmin (dalteparin sodium) as part of routine clinical practice and is expected to be treated conservatively (without PCI or CABG within 48 hours) during the index hospitalization.
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Patients who are contraindicated to receive this agent per the local approved prescribing information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients management of non-ST segment elevated acute coronary syndromes in nursing home who will be treated conservatively (without percutaneous corornary intervention [PCI] or coronary artery bypass graft [CABG] within 48 hours).
Sampling Method: Non-Probability Sample
Enrollment: 618 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- India (17):
  - Pfizer Investigational Site, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Surat, Gujarat
  - Pfizer Investigational Site, Hisar, Haryana
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Manglore, Karnataka
  - Pfizer Investigational Site, Mysore, Karnataka
  - Pfizer Investigational Site, Nagpur, Maharahtra
  - Pfizer Investigational Site, Nashik, Maharahtra
  - Pfizer Investigational Site, Ambernath (E), Maharashtra
  - Pfizer Investigational Site, Nagpur, Maharashtra
  - Pfizer Investigational Site, Nashik, Maharashtra
  - Pfizer Investigational Site, Nashik Road, Maharashtra
  - Pfizer Investigational Site, Thane, Maharashtra
  - Pfizer Investigational Site, Bikaner, Rajasthan
  - Pfizer Investigational Site, Jaipur, Rajasthan
  - Pfizer Investigational Site, Chennai, Tamil Nadu
  - Pfizer Investigational Site, Kolkata, West Bengal

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6301088&StudyName=Effectiveness%20And%20Safety%20Of%20Dalteparin%20In%20Patients%20With%20Acute%20Coronary%20Syndromes%20Without%20ST%20Elevations%20In%20Clinical%20Practice

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 618 participants were screened, of which 617 participant were assigned to study treatment and 1 participant was excluded based on investigator's discretion.
Groups:
- Dalteparin: Dalteparin Sodium 120 international units/kilogram (IU/kg) total body weight up to a maximum dose of 10,000 IU subcutaneously (s.c.) every 12 hours, for 1-2 weeks.
Period: Overall Study
Arm/Group | Dalteparin
Started | 617
Completed | 610
Not Completed | 7
Not completed — Death | 3
Not completed — Withdrawal by Subject | 2
Not completed — Other | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dalteparin
Number analyzed (Participants) | 617
Age Continuous [Mean (Standard Deviation); unit: years] | 57.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 249
  Male | 368

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Death or Myocardial Infarction (MI)
Time Frame: Baseline to 28 days after last dose of study drug
Population: The full analysis set (FAS) included all enrolled participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Dalteparin
Number analyzed (Participants) | 617
Participants | 3

2. Primary Outcome: Number of Participants With Major Bleeding Events
Description: Bleeding events were considered major if, accompanied by a decrease in hemoglobin of more than or equal to 2 grams/deciliter (g/dL) in connection with clinical symptoms; a transfusion was required; bleeding led to interruption of treatment or death; or intracranial bleeding.
Time Frame: Baseline to 28 days after last dose of study drug
Population: FAS included all enrolled participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Dalteparin
Number analyzed (Participants) | 617
Participants | 0

3. Primary Outcome: Number of Participants With Minor Bleeding Events
Description: Bleeding events like hematuria, wound hematoma or injection site hematoma which did not fulfill the criteria for a major bleeding episode were classified as minor bleeding.
Time Frame: Baseline to 28 days after last dose of study drug
Population: FAS included all enrolled participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Dalteparin
Number analyzed (Participants) | 617
Participants | 1

4. Other Pre Specified Outcome: Number of Participants With Stroke
Description: Stroke was defined as a sudden, focal neurologic deficit that was not reversible within 24 hours and was not the result of any readily identifiable cause (for example, tumor or trauma).
Time Frame: Baseline to 28 days after last dose of study drug
Population: FAS included all enrolled participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Dalteparin
Number analyzed (Participants) | 617
Participants | 0

5. Other Pre Specified Outcome: Number of Participants With Cardiac Arrest- Resuscitated
Description: Cardiac arrest resuscitated was defined as sudden cessation of cardiac activity so that the participant became unresponsive, with no normal breathing and no signs of circulation. Cardiac arrest was used to signify an event that was reversed, usually by cardio-pulmonary resuscitation (CPR) and/or defibrillation or cardioversion, or cardiac pacing.
Time Frame: Baseline to 28 days after last dose of study drug
Population: FAS included all enrolled participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Dalteparin
Number analyzed (Participants) | 617
Participants | 2

6. Other Pre Specified Outcome: Number of Participants With Heparin Induced Thrombocytopenia
Description: Thrombocytopenia was defined as a disorder in which there is an abnormally low platelet count. A normal platelet count ranged from 150,000 to 450,000 platelets per micro liter of blood.
Time Frame: Baseline to 28 days after last dose of study drug
Population: FAS included all enrolled participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Dalteparin
Number analyzed (Participants) | 617
Participants | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Dalteparin
Serious Adverse Events (participants affected / at risk) | 4/617
Other Adverse Events (participants affected / at risk) | 23/617
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalteparin (N=617)
Cardiac Arrest (Cardiac disorders) | 2
Cardio-respiratory Arrest (Cardiac disorders) | 2
Left Ventricular Failure (Cardiac disorders) | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalteparin (N=617)
Anaemia (Blood and lymphatic system disorders) | 3
Abdominal Pain (Gastrointestinal disorders) | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 1
Gingival Bleeding (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest Pain (General disorders) | 2
Chills (General disorders) | 1
Pyrexia (General disorders) | 3
Hepatitis (Hepatobiliary disorders) | 1
Lower Respiratory Tract Infections (Infections and infestations) | 1
Respiratory Rate (Investigations) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 3
Hemiplegia (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1
Venous Thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.